CLINICAL TRIAL: NCT02879318
Title: A Randomized Phase II Trial of Gemcitabine and Nab-Paclitaxel vs Gemcitabine, Nab-Paclitaxel, Durvalumab and Tremelimumab as 1st Line Therapy in Metastatic Pancreatic Adenocarcinoma
Brief Title: Gemcitabine and Nab-Paclitaxel vs Gemcitabine, Nab-Paclitaxel, Durvalumab and Tremelimumab as 1st Line Therapy in Metastatic Pancreatic Adenocarcinoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Canadian Cancer Trials Group (Network)
Collaborators: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PA7
Record Dates: First submitted 2016-08-22; First posted 2016-08-25 (Estimated); Results first posted 2021-05-28 (Actual); Last update posted 2025-03-24 (Actual); Status verified 2025-03

CONDITIONS: Pancreatic Adenocarcinoma
MeSH Terms: interventions — Gemcitabine; 130-nm albumin-bound paclitaxel; durvalumab; tremelimumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Gemcitabine plus Nab-Paclitaxel (Active Comparator): Gemcitabine 1000 mg/m2 IV & Nab-Paclitaxel 125 mg/m2 until unequivocal progression or unacceptable toxicity. Days 1, 8, 15 Q28 days.
  Interventions: Drug: Gemcitabine; Drug: Nab-paclitaxel
- Gemcitabine + Nab-Paclitaxel + Durvalumab + Tremelimumab (Experimental): Gemcitabine 1000 mg/m2 IV & Nab-Paclitaxel 125 mg/m2 until unequivocal progression or unacceptable toxicity. Day 1, 8, 15 Q28 days.
  plus Durvalumab 1500mg IV day 1 only Q28 days; and Tremelimumab 75 mg IV Days 1 cycles 1, 2, 3 and 4 only until unequivocal progression or unacceptable toxicity.
  Interventions: Drug: Gemcitabine; Drug: Nab-paclitaxel; Drug: Durvalumab; Drug: Tremelimumab

INTERVENTIONS:
Drug: Gemcitabine
Drug: Nab-paclitaxel
Drug: Durvalumab
  Arms: Gemcitabine + Nab-Paclitaxel + Durvalumab + Tremelimumab
Drug: Tremelimumab
  Arms: Gemcitabine + Nab-Paclitaxel + Durvalumab + Tremelimumab

SUMMARY:
The standard or usual treatment for this disease consists of two chemotherapy drugs gemcitabine and nab-paclitaxel given together.

DETAILED DESCRIPTION:
Durvalumab is a new type of drug for many types of cancer. Laboratory tests show that it works by allowing the immune system to detect cancer and reactivate the immune response. This may halp to slow down the growth of cancer or may cause cancer cells to die. Durvalumab has been shown to shrink tumours in animals and has been studied in a few people and seems promising but it is not clear if it can offer better results than standard treatments alone.

Tremelimumab is a new type of drug for various types of cancers. It works in a similar way to durvalumab and may improve the effect of durvalumab. This may also help slow the growth of the cancer cells or may cause cancer cells to die. Tremelimumab has been shown to shrink tumours in animals and has been studied in a few people and seems promising but it is not clear if it can offer better results than standard treatment alone when used with durvalumab.

Combination of durvalumab and tremelimumab have also been studied and when combined have been shown to increase tumour shrinkage in animals compared to either drug alone and while the combination has been studied in a few people, it is not clear if it can offer better results than standard treatment.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically or cytologically confirmed pancreatic ductal adenocarcinoma which is metastatic.
* Must have presence of measurable or evaluable disease as defined by Response Evaluation Criteria in Solid Tumours (RECIST 1.1).
* Patients must be considered suitable candidates for, and able to receive, first line chemotherapy for metastatic disease with gemcitabine and nab-paclitaxel.
* Patient must consent to provision of, and investigator(s) must confirm access to and agree to submit within 4 weeks of randomization to the CCTG Central Tumour Bank, a representative formalin fixed paraffin block of tumour tissue of adequate amount and quality in order that the specific correlative marker assays proscribed in the protocol may be conducted.
* Patient must consent to provision of samples of blood, serum and plasma in order that the specific correlative marker assays proscribed may be conducted.
* Patients must be ≥ 18 years of age.
* Patients must have an ECOG performance status of 0 or 1 with a life expectancy of at least 12 weeks.
* No prior treatment for metastatic disease is permitted. Patients may have received prior adjuvant chemotherapy if the last dose was given more than 6 months prior to recurrence. Patients may not have received chemoradiotherapy or adjuvant radiation therapy. Patient may not have received nab-paclitaxel as adjuvant therapy. Prior systemic treatment for borderline resectable or locally advanced disease is not permitted. Patients receiving a single dose of radiation (up to 8Gy/800RAD) with palliative intent for pain control are eligible provided a minimum of 14 days have elapsed between the radiation and the date of randomization.
* Adequate normal organ and marrow function as defined below (must be done within 14 days prior to registration).

Absolute neutrophils ≥ 1.5 x 10^9/L Platelets ≥ 100 x 10^9/L Hemoglobin ≥90 g/L Bilirubin ≤ 1.5 x upper normal limit AST and ALT ≤ 2.5 x upper normal limit Serum creatinine <1.25 UNL or Creatinine clearance ≥40mL/min

* Imaging investigations including CT/MRI of chest/abdomen/pelvis or other scans as necessary to document all sites of disease done within 28 days prior to randomization.
* Patient is able (i.e. sufficiently fluent) and willing to complete the quality of life questionnaires in either English or French.
* Patient consent must be appropriately obtained in accordance with applicable local and regulatory requirements.
* Patients must be accessible for treatment and follow-up. Patients registered on this trial must be treated and followed at the participating centre. Patients must agree to return to the participating centre for management of any adverse events which may occur through the course of the trial. This implies there must be reasonable geographical limits placed on patients being considered for this trial. Sites are encouraged to contact CCTG (or their respective Cooperative Group for sites outside Canada) for any questions regarding the interpretation of this criterion. Investigators must assure themselves the patients randomized on this trial will be available for complete documentation of the treatment, adverse events, and follow-up.
* In accordance with CCTG policy, protocol treatment is to begin within 2 working days of patient randomization.
* Women/men of childbearing potential must have agreed to use a highly effective contraceptive method

Exclusion Criteria:

* Patients with a history of other malignancies, except: adequately treated non-melanoma skin cancer, curatively treated in-situ cancer of the cervix, or other solid tumours curatively treated with no evidence of disease for ≥ 5 years. Patients with a history of other malignancies detected at an early stage and whom the investigator believes have been curatively treated and are at a low risk of recurrence MAY be eligible. Contact CCTG to discuss eligibility prior to enrolling.
* Any previous treatment with a PD1 or PD-L1 inhibitor, including durvalumab or an anti-CTLA4, including tremelimumab.
* History of primary immunodeficiency, history of organ transplant that requires therapeutic immunosuppression or prior history of severe (grade 3 or 4) immune-mediated toxicity from other immune therapy.
* Current or prior use of immunosuppressive medication within 28 days before the first planned dose of study therapy, with the exceptions of intranasal and inhaled corticosteroids or systemic corticosteroids at physiological doses, which are not to exceed 10 mg/day of prednisone, or an equivalent corticosteroid.
* Active or prior documented autoimmune or inflammatory disorders (including inflammatory bowel disease (e.g. colitis or Crohn's disease) diverticulitis with the exception of diverticulosis, celiac disease or other serious gastrointestinal chronic conditions associated with diarrhea), systemic lupus erythematosus, Sarcoidosis syndrome, or Wegener syndrome (granulomatosis with polyangitis), rheumatoid arthritis, hypophysitis, uveitis, etc. within the past 3 years prior to the start of treatment. The following are exceptions to this criterion:

  * Patients with alopecia
  * Patients with Grave's disease, vitiligo or psoriasis not requiring systemic treatment (within the last 2 years).
  * Patients with hypothyroidism (e.g. following Hashimoto syndrome) stable on hormone replacement.

NOTE: Patients with vitiligo, Grave's disease, or psoriasis not requiring systemic treatment (within the past 2 years) are not excluded.

* Patients with active or uncontrolled intercurrent illness including, but not limited to:

  * cardiac dysfunction (symptomatic congestive heart failure, uncontrolled hypertension, unstable angina pectoris, cardiac arrhythmia);
  * active peptic ulcer disease or gastritis;
  * active bleeding diatheses;
  * psychiatric illness/social situations that would limit compliance with study requirements or compromise the ability of the subject to give written informed consent;
  * known history of previous clinical diagnosis of tuberculosis;
  * known human immunodeficiency virus infection (positive HIV 1/2 antibodies);
  * known active hepatitis B infection (positive HBV surface antigen (HBsAg)). Patients with a past or resolved HBV infection (defined as presence of hepatitis B core antibody (anti-HBc) and absence of HBsAg) are eligible;
  * known active hepatitis C infection. Patients positive for hepatitis C (HCV) antibody are eligible only if polymerase chain reaction is negative for HCV RNA.
* History of leptomeningeal carcinomatosis.
* Symptomatic or uncontrolled brain metastases requiring concurrent treatment, inclusive of but not limited to surgery, radiation and/or corticosteroids.
* Receipt of live attenuated vaccination (examples include, but are not limited to, vaccines for measles, mumps, and rubella, live attenuated influenza vaccine (nasal), chicken pox vaccine, oral polio vaccine, rotavirus vaccine, yellow fever vaccine, BCG vaccine, typhoid vaccine and typhus vaccine) within 30 days prior to randomization.
* Pregnant or lactating women.
* Any active disease condition which would render the protocol treatment dangerous or impair the ability of the patient to receive protocol therapy.
* Any condition (e.g. psychological, geographical, etc.) that does not permit compliance with the protocol.
* History of hypersensitivity to gemcitabine, nab-paclitaxel, durvalumab or tremelimumab or any excipient.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Actual)
Dates: Start 2016-11-07 (Actual); Primary Completion 2020-08-03 (Actual); Study Completion 2025-03-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Derek Jonker, Study Chair — Ottawa Hospital Research Institute, ON Canada
Locations (27):
- Canada (27):
  - Tom Baker Cancer Centre, Calgary, Alberta
  - BCCA - Vancouver Cancer Centre, Vancouver, British Columbia
  - CancerCare Manitoba, Winnipeg, Manitoba
  - The Moncton Hospital, Moncton, New Brunswick
  - The Vitalite Health Network - Dr. Leon Richard, Moncton, New Brunswick
  - Dr. H. Bliss Murphy Cancer Centre, St. John's, Newfoundland and Labrador
  - QEII Health Sciences Centre, Halifax, Nova Scotia
  - Juravinski Cancer Centre at Hamilton Health Sciences, Hamilton, Ontario
  - Kingston Health Sciences Centre, Kingston, Ontario
  - Grand River Regional Cancer Centre, Kitchener, Ontario
  - London Regional Cancer Program, London, Ontario
  - Ottawa Hospital Research Institute, Ottawa, Ontario
  - Algoma District Cancer Program, Sault Ste. Marie, Ontario
  - Niagara Health System, St. Catharines, Ontario
  - Odette Cancer Centre, Toronto, Ontario
  - University Health Network, Toronto, Ontario
  - St. Joseph's Health Centre, Toronto, Ontario
  - Hopital de la Cite-de-la-Sante, Laval, Quebec
  - L'Hotel-Dieu de Levis, Lévis, Quebec
  - CHUM-Centre Hospitalier de l'Universite de Montreal, Montreal, Quebec
  - The Jewish General Hospital, Montreal, Quebec
  - The Research Institute of the McGill University, Montreal, Quebec
  - Centre Integre Universitaire De Sante Et De Services, Montreal, Quebec
  - CHUQ-Pavillon Hotel-Dieu de Quebec, Québec, Quebec
  - Centre hospitalier universitaire de Sherbrooke, Sherbrooke, Quebec
  - Allan Blair Cancer Centre, Regina, Saskatchewan
  - Saskatoon Cancer Centre, Saskatoon, Saskatchewan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Renouf DJ, Loree JM, Knox JJ, Topham JT, Kavan P, Jonker D, Welch S, Couture F, Lemay F, Tehfe M, Harb M, Aucoin N, Ko YJ, Tang PA, Ramjeesingh R, Meyers BM, Kim CA, Du P, Jia S, Schaeffer DF, Gill S, Tu D, O'Callaghan CJ. The CCTG PA.7 phase II trial of gemcitabine and nab-paclitaxel with or without durvalumab and tremelimumab as initial therapy in metastatic pancreatic ductal adenocarcinoma. Nat Commun. 2022 Aug 26;13(1):5020. doi: 10.1038/s41467-022-32591-8. PMID 36028483

RESULTS

PARTICIPANT FLOW:
Recruitment Details: From April 10, 2017 to July 28, 2018 in 25 cancer centres in Canada
Pre-assignment Details: There was a run-in phase of this study which accrued the first patient on August 22, 2016, which can be considered as start date of this study. Only patients recruited from April 10, 2017 to July 28, 2018 into the randomized phase II component of the study were included in the analysis.
Groups:
- Gemcitabine Plus Nab-Paclitaxel: Gemcitabine 1000 mg/m2 IV & Nab-Paclitaxel 125 mg/m2 until unequivocal progression or unacceptable toxicity. Days 1, 8, 15 Q28 days.
  Gemcitabine
  Nab-paclitaxel
- Gemcitabine + Nab-Paclitaxel + Durvalumab + Tremelimumab: Gemcitabine 1000 mg/m2 IV & Nab-Paclitaxel 125 mg/m2 until unequivocal progression or unacceptable toxicity. Day 1, 8, 15 Q28 days.
  plus Durvalumab 1500mg IV day 1 only Q28 days; and Tremelimumab 75 mg IV Days 1 cycles 1, 2, 3 and 4 only until unequivocal progression or unacceptable toxicity.
  Gemcitabine
  Nab-paclitaxel
  Durvalumab
  Tremelimumab
Period: Overall Study
Arm/Group | Gemcitabine Plus Nab-Paclitaxel | Gemcitabine + Nab-Paclitaxel + Durvalumab + Tremelimumab
Started | 61 | 119
Completed | 61 | 119
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Gemcitabine Plus Nab-Paclitaxel | Gemcitabine + Nab-Paclitaxel + Durvalumab + Tremelimumab | Total
Number analyzed (Participants) | 61 | 119 | 180
Age, Continuous [Median (Full Range); unit: years] | 65 [42 to 84] | 64 [29 to 81] | 65 [29 to 84]
Age, Customized [Count of Participants; unit: Participants]
  Younger than 65 years | 27 | 61 | 88
  65 years or older | 34 | 58 | 92
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 35 | 52 | 87
  Male | 26 | 67 | 93
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 6 | 10 | 16
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 2 | 2
  White | 55 | 105 | 160
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 2 | 2
Region of Enrollment [Number; unit: participants]
  Canada | 61 | 119 | 180
Eastern Cooperative Oncology Group (ECOG) Performance Status [Count of Participants; unit: Participants] — 0: Fully active, able to carry on all pre-disease performance without restriction
  1. Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature, e.g., light house work, office work
  2. Ambulatory and capable of all selfcare but unable to carry out any work activities; up and about more than 50% of waking hours
  3. Capable of only limited selfcare; confined to bed or chair more than 50% of waking hours
  4. Completely disabled; cannot carry on any selfcare; totally confined to bed or chair 5. Dead
  Participants
    0 | 14 | 27 | 41
    1 | 47 | 92 | 139

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival
Description: Time from randomization to death from any cause with patients who were alive at the time of the final analysis or who became lost to follow-up censored at their last date known to be alive.
Time Frame: 35 months
Measure: Median (90% Confidence Interval); unit: months
Arm/Group | Gemcitabine Plus Nab-Paclitaxel | Gemcitabine + Nab-Paclitaxel + Durvalumab + Tremelimumab
Number analyzed (Participants) | 61 | 119
months | 8.8 [7.2 to 11.2] | 9.8 [8.3 to 12.2]
Statistical Analysis 1: Comparison: Gemcitabine Plus Nab-Paclitaxel vs Gemcitabine + Nab-Paclitaxel + Durvalumab + Tremelimumab; Test type: Superiority; p = 0.72, Log Rank — a priori threshold for statistical significance was 0.1; stratified by ECOG performance status and prior adjuvant therapy; Hazard Ratio (HR) = 0.94, 90% CI 2-sided [0.71 to 1.25]

2. Secondary Outcome: Progression Free Survival
Description: Defined as the time from randomization to the first objective documentation of disease progression, defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0), as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions, or death due to any cause with patients who had not progressed or died at the time of final analysis censored on the date of the last tumour assessment.
Time Frame: 35 months
Measure: Median (90% Confidence Interval); unit: months
Arm/Group | Gemcitabine Plus Nab-Paclitaxel | Gemcitabine + Nab-Paclitaxel + Durvalumab + Tremelimumab
Number analyzed (Participants) | 61 | 119
months | 5.4 [3.6 to 6.6] | 5.5 [3.8 to 5.7]
Statistical Analysis 1: Comparison: Gemcitabine Plus Nab-Paclitaxel vs Gemcitabine + Nab-Paclitaxel + Durvalumab + Tremelimumab; Test type: Superiority; p = 0.91, Log Rank; Hazard Ratio (HR) = 0.98, 90% CI 2-sided [0.75 to 1.29]

3. Secondary Outcome: Objective Response Rate
Description: Defined as percentage of participants with objective response over all participants randomized. Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0) for target lesions and assessed by MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Objective Response (OR) = CR + PR.
Time Frame: 35 months
Measure: Count of Participants; unit: Participants
Arm/Group | Gemcitabine Plus Nab-Paclitaxel | Gemcitabine + Nab-Paclitaxel + Durvalumab + Tremelimumab
Number analyzed (Participants) | 61 | 119
Participants
  Responded | 14 | 36
  Not responded | 47 | 83
Statistical Analysis 1: Comparison: Gemcitabine Plus Nab-Paclitaxel vs Gemcitabine + Nab-Paclitaxel + Durvalumab + Tremelimumab; Test type: Superiority; p = 0.28, Cochran-Mantel-Haenszel; stratified by ECOG performance status and prior adjuvant chemotherapy; Odds Ratio (OR) = 1.49, 90% CI 2-sided [0.81 to 2.72]

ADVERSE EVENTS:
Time Frame: 35 months
Description: Only patients who received at least one dose of protocol treatment were included in the evaluation of adverse events.
Arm/Group | Gemcitabine Plus Nab-Paclitaxel | Gemcitabine + Nab-Paclitaxel + Durvalumab + Tremelimumab
All-Cause Mortality (participants affected / at risk) | 52/58 | 102/119
Serious Adverse Events (participants affected / at risk) | 26/58 | 82/119
Other Adverse Events (participants affected / at risk) | 57/58 | 118/119
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Gemcitabine Plus Nab-Paclitaxel (N=58) | Gemcitabine + Nab-Paclitaxel + Durvalumab + Tremelimumab (N=119)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 | 6
Leukocytosis (Blood and lymphatic system disorders) | 0 | 1
Cardiac arrest (Cardiac disorders) | 0 | 2
Heart failure (Cardiac disorders) | 1 | 0
Myocarditis (Cardiac disorders) | 0 | 1
Pericardial effusion (Cardiac disorders) | 0 | 1
Abdominal distension (Gastrointestinal disorders) | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 6 | 5
Colitis (Gastrointestinal disorders) | 0 | 5
Colonic obstruction (Gastrointestinal disorders) | 0 | 1
Colonic perforation (Gastrointestinal disorders) | 0 | 1
Constipation (Gastrointestinal disorders) | 1 | 1
Diarrhea (Gastrointestinal disorders) | 1 | 3
Duodenal obstruction (Gastrointestinal disorders) | 0 | 1
Duodenal stenosis (Gastrointestinal disorders) | 0 | 2
Enterocolitis (Gastrointestinal disorders) | 0 | 1
Gastric hemorrhage (Gastrointestinal disorders) | 1 | 1
Gastric ulcer (Gastrointestinal disorders) | 1 | 0
Gastrointestinal pain (Gastrointestinal disorders) | 0 | 1
Ileal obstruction (Gastrointestinal disorders) | 0 | 1
Ileus (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 1 | 2
Obstruction gastric (Gastrointestinal disorders) | 1 | 1
Other gastrointestinal disorders (Gastrointestinal disorders) | 0 | 1
Pancreatic duct stenosis (Gastrointestinal disorders) | 0 | 1
Pancreatitis (Gastrointestinal disorders) | 1 | 1
Proctitis (Gastrointestinal disorders) | 0 | 1
Small intestinal obstruction (Gastrointestinal disorders) | 1 | 2
Small intestinal perforation (Gastrointestinal disorders) | 0 | 1
Upper gastrointestinal hemorrhage (Gastrointestinal disorders) | 0 | 2
Vomiting (Gastrointestinal disorders) | 1 | 5
Chills (General disorders) | 0 | 1
Death NOS (General disorders) | 1 | 0
Edema limbs (General disorders) | 1 | 3
Edema trunk (General disorders) | 0 | 1
Fatigue (General disorders) | 1 | 5
Fever (General disorders) | 4 | 14
Sudden death NOS (General disorders) | 0 | 1
Bile duct stenosis (Hepatobiliary disorders) | 0 | 6
Gallbladder obstruction (Hepatobiliary disorders) | 0 | 1
Hepatic failure (Hepatobiliary disorders) | 0 | 1
Other immune system disorders (Immune system disorders) | 0 | 8
Appendicitis (Infections and infestations) | 0 | 1
Biliary tract infection (Infections and infestations) | 3 | 10
Catheter related infection (Infections and infestations) | 1 | 0
Enterocolitis infectious (Infections and infestations) | 1 | 1
Hepatic infection (Infections and infestations) | 0 | 3
Lung infection (Infections and infestations) | 2 | 5
Other infections and infestations (Infections and infestations) | 0 | 1
Sepsis (Infections and infestations) | 7 | 12
Skin infection (Infections and infestations) | 0 | 1
Upper respiratory infection (Infections and infestations) | 0 | 2
Urinary tract infection (Infections and infestations) | 0 | 2
Aortic injury (Injury, poisoning and procedural complications) | 0 | 1
Fall (Injury, poisoning and procedural complications) | 0 | 1
Hip fracture (Injury, poisoning and procedural complications) | 1 | 0
Spinal fracture (Injury, poisoning and procedural complications) | 1 | 1
Blood bilirubin increased (Investigations) | 0 | 1
Platelet count decreased (Investigations) | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 4
Hypercalcemia (Metabolism and nutrition disorders) | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 2
Bone pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 2 | 1
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 0 | 1
Encephalopathy (Nervous system disorders) | 0 | 1
Ischemia cerebrovascular (Nervous system disorders) | 0 | 1
Lethargy (Nervous system disorders) | 0 | 1
Presyncope (Nervous system disorders) | 0 | 2
Radiculitis (Nervous system disorders) | 0 | 1
Reversible posterior leukoencephalopathy syndrome (Nervous system disorders) | 0 | 1
Stroke (Nervous system disorders) | 0 | 3
Confusion (Psychiatric disorders) | 1 | 1
Delirium (Psychiatric disorders) | 0 | 2
Insomnia (Psychiatric disorders) | 0 | 1
Acute kidney injury (Renal and urinary disorders) | 1 | 2
Urinary tract obstruction (Renal and urinary disorders) | 0 | 1
Adult respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 | 9
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 3
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 | 7
Pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Photosensitivity (Skin and subcutaneous tissue disorders) | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 2
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 4
Skin ulceration (Skin and subcutaneous tissue disorders) | 0 | 1
Hypertension (Vascular disorders) | 0 | 1
Hypotension (Vascular disorders) | 1 | 4
Other vascular disorders (Vascular disorders) | 0 | 1
Superficial thrombophlebitis (Vascular disorders) | 0 | 1
Thromboembolic event (Vascular disorders) | 1 | 5
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Gemcitabine Plus Nab-Paclitaxel (N=58) | Gemcitabine + Nab-Paclitaxel + Durvalumab + Tremelimumab (N=119)
Hearing impaired (Ear and labyrinth disorders) | 3 | 3
Blurred vision (Eye disorders) | 2 | 12
Dry eye (Eye disorders) | 3 | 7
Abdominal distension (Gastrointestinal disorders) | 4 | 10
Abdominal pain (Gastrointestinal disorders) | 45 | 93
Ascites (Gastrointestinal disorders) | 3 | 5
Bloating (Gastrointestinal disorders) | 2 | 14
Constipation (Gastrointestinal disorders) | 33 | 80
Diarrhea (Gastrointestinal disorders) | 33 | 76
Dry mouth (Gastrointestinal disorders) | 5 | 9
Dyspepsia (Gastrointestinal disorders) | 9 | 20
Flatulence (Gastrointestinal disorders) | 1 | 6
Gastroesophageal reflux disease (Gastrointestinal disorders) | 10 | 17
Gastrointestinal pain (Gastrointestinal disorders) | 1 | 6
Hemorrhoidal hemorrhage (Gastrointestinal disorders) | 3 | 0
Hemorrhoids (Gastrointestinal disorders) | 1 | 8
Mucositis oral (Gastrointestinal disorders) | 4 | 12
Nausea (Gastrointestinal disorders) | 41 | 88
Other gastrointestinal disorders (Gastrointestinal disorders) | 0 | 6
Stomach pain (Gastrointestinal disorders) | 2 | 12
Vomiting (Gastrointestinal disorders) | 28 | 60
Chills (General disorders) | 6 | 19
Edema face (General disorders) | 1 | 6
Edema limbs (General disorders) | 25 | 57
Fatigue (General disorders) | 48 | 103
Fever (General disorders) | 18 | 48
Flu like symptoms (General disorders) | 5 | 15
Non-cardiac chest pain (General disorders) | 0 | 19
Pain (General disorders) | 4 | 11
Lung infection (Infections and infestations) | 4 | 12
Mucosal infection (Infections and infestations) | 0 | 7
Skin infection (Infections and infestations) | 8 | 16
Upper respiratory infection (Infections and infestations) | 5 | 7
Urinary tract infection (Infections and infestations) | 7 | 9
Bruising (Injury, poisoning and procedural complications) | 4 | 4
Fall (Injury, poisoning and procedural complications) | 3 | 5
Wound complication (Injury, poisoning and procedural complications) | 3 | 1
Weight loss (Investigations) | 17 | 31
Anorexia (Metabolism and nutrition disorders) | 35 | 76
Dehydration (Metabolism and nutrition disorders) | 6 | 15
Arthralgia (Musculoskeletal and connective tissue disorders) | 6 | 28
Back pain (Musculoskeletal and connective tissue disorders) | 23 | 62
Bone pain (Musculoskeletal and connective tissue disorders) | 4 | 5
Flank pain (Musculoskeletal and connective tissue disorders) | 4 | 7
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 7 | 16
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 4 | 7
Myalgia (Musculoskeletal and connective tissue disorders) | 3 | 17
Pain in extremity (Musculoskeletal and connective tissue disorders) | 7 | 27
Dizziness (Nervous system disorders) | 9 | 24
Dysgeusia (Nervous system disorders) | 16 | 34
Headache (Nervous system disorders) | 13 | 26
Paresthesia (Nervous system disorders) | 7 | 17
Peripheral motor neuropathy (Nervous system disorders) | 6 | 9
Peripheral sensory neuropathy (Nervous system disorders) | 20 | 59
Somnolence (Nervous system disorders) | 0 | 6
Anxiety (Psychiatric disorders) | 9 | 33
Confusion (Psychiatric disorders) | 2 | 8
Depression (Psychiatric disorders) | 5 | 17
Insomnia (Psychiatric disorders) | 17 | 53
Libido decreased (Psychiatric disorders) | 3 | 0
Hematuria (Renal and urinary disorders) | 0 | 7
Urinary frequency (Renal and urinary disorders) | 5 | 6
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 5 | 12
Cough (Respiratory, thoracic and mediastinal disorders) | 14 | 35
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 22 | 56
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 12 | 22
Hiccups (Respiratory, thoracic and mediastinal disorders) | 2 | 6
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 3 | 9
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 5 | 7
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 3 | 6
Productive cough (Respiratory, thoracic and mediastinal disorders) | 5 | 6
Sore throat (Respiratory, thoracic and mediastinal disorders) | 3 | 11
Alopecia (Skin and subcutaneous tissue disorders) | 28 | 64
Dry skin (Skin and subcutaneous tissue disorders) | 5 | 17
Erythema multiforme (Skin and subcutaneous tissue disorders) | 1 | 6
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 | 13
Nail discoloration (Skin and subcutaneous tissue disorders) | 1 | 8
Other skin and subcutaneous tissue disorders (Skin and subcutaneous tissue disorders) | 1 | 10
Pain of skin (Skin and subcutaneous tissue disorders) | 2 | 7
Pruritus (Skin and subcutaneous tissue disorders) | 6 | 29
Rash acneiform (Skin and subcutaneous tissue disorders) | 3 | 15
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 14 | 51
Hot flashes (Vascular disorders) | 2 | 9
Hypertension (Vascular disorders) | 7 | 11
Hypotension (Vascular disorders) | 4 | 9
Thromboembolic event (Vascular disorders) | 17 | 30

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2018-03-20): https://cdn.clinicaltrials.gov/large-docs/18/NCT02879318/Prot_000.pdf
  • Statistical Analysis Plan (2019-08-09): https://cdn.clinicaltrials.gov/large-docs/18/NCT02879318/SAP_001.pdf